CLINICAL TRIAL: NCT01292239
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Trial in Japan to Investigate the Efficacy and Safety of TMC435 vs. Placebo as Part of a Treatment Regimen Including Peginterferon Alfa-2a and Ribavirin in Treatment-Naive, Genotype 1, Hepatitis C-infected Subjects
Brief Title: A Phase III Study of TMC435 in Treatment-naive, Genotype 1, Hepatitis C-infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR017686; TMC435HPC3003 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-02-01; First posted 2011-02-09 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Hepatitis C; Hepatitis C virus; Interferon Alfa-2a; Ribavirin; Viral RNA
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMC435 100 mg 12 Wks + PR 24/48 (Experimental): Participants received TMC435 100 mg once daily with PegIFNα-2a and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 24. Treatment was stopped at Week 24 for participants who achieved HCV RNA < 1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable HCV RNA at Week 12. All other participants continued PR until Week 48.
  Interventions: Drug: TMC435; Drug: Peginterferon alfa-2a (pegIFN alfa-2a); Drug: Ribavirin (RBV)
- PBO 12 Wks + PR 48 (Experimental): Participants received placebo (PBO) once daily with PegIFNα-2a and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 48.
  Interventions: Drug: Placebo; Drug: Peginterferon alfa-2a (pegIFN alfa-2a); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Placebo — Placebo capsule taken by mouth once daily for 12 weeks
  Arms: PBO 12 Wks + PR 48
Drug: TMC435 — 100-mg capsule taken by mouth once daily for 12 weeks
  Arms: TMC435 100 mg 12 Wks + PR 24/48
Drug: Peginterferon alfa-2a (pegIFN alfa-2a) — PegIFN alfa-2a (PEGASYS) will be administered according to the manufacturer's prescribing information as 180 mcg once weekly injected subcutaneous (under the skin) for up to 24-48 weeks for patients randomized to TMC435 and for up to 48 weeks for patients randomized to placebo.
  Other Names: PEGASYS
Drug: Ribavirin (RBV) — RBV (COPEGUS) will be administered according to the manufacturer's prescribing information. If body weight is > 80 kg the total daily dose of RBV will be 1000 mg, taken by mouth as 400 mg (2 tablets of 200 mg) after breakfast and 600 mg (3 tablets of 200 mg) after supper. If body weight is > 60 kg to <=80 kg the total daily dose will be 800 mg, taken by mouth as 400 mg (2 tablets of 200 mg per intake) after breakfast and supper. If body weight is <=60 kg the total daily dose of RBV will be 600 mg, taken by mouth as 200 mg (1 tablet of 200 mg) after breakfast and 400 mg (2 tablets of 200 mg) after supper. Total duration of RBV will be 24-48 weeks.
  Other Names: COPEGUS

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TMC435 compared with placebo in combination with peginterferon alfa-2a (pegIFN alfa-2a) and ribavirin in treatment-naive patients with chronic genotype 1 hepatitis C virus (HCV) infection in Japan.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), 2-arm, double-blind study to evaluate the efficacy and safety of TMC435 (also referred to as jnj-38733214-aaa) versus placebo in combination with the standard of care (SoC) therapy (peginterferon alfa-2a [pegIFN alfa-2a] and ribavirin) in adult treatment-naïve patients (who never received treatment for HCV) with chronic genotype 1 HCV infection in Japan. The study objective is to evaluate and compare the efficacy of TMC435 vs placebo by the proportion of the patients with undetectable HCV ribonucleic acid (RNA). In the TMC435 treatment group, patients will receive 12 weeks of treatment with TMC435 (100 mg) once daily plus SoC followed by an additional 12 or 36 weeks of treatment with SoC. In the placebo treatment group, patients will receive 12 weeks of treatment with placebo once daily plus SoC followed by an additional 36 weeks of treatment with SoC. TMC435 is a 100-mg capsule and will be taken orally by mouth. The SoC treatment will be given for 24 or 48 weeks. Pegylated interferon is supplied as a vial containing 1.0 mL solution with 180 mcg pegIFN alpha-2a and administered subcutaneously (injected by a syringe under the skin) once weekly. Ribavirin is given as 200-mg tablets (daily dose: 600-1000 mg based on body weight), and taken orally by mouth two times a day after meals.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have chronic genotype 1 HCV infection with HCV RNA level >= 5.0 log10 IU/mL
* Patient has never received treatment for HCV
* Patient must be willing to use contraceptive measures from the time of informed consent to 6 months after last dose of study medication

Exclusion Criteria:

* Co-infection with any other HCV genotype or co-infection with the human immunodeficiency virus (HIV)
* Diagnosed with hepatic cirrhosis or hepatic failure
* A medical condition which is a contraindication to pegIFN or ribavirin therapy
* History of, or any current medical condition which could impact the safety of the patient in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (28):
- Japan (28):
  - Amagasaki
  - Chiba
  - Chūō
  - Hiroshima
  - Ichikawa
  - Ikeda
  - Inashiki
  - Iruma
  - Kagoshima
  - Kanazawa
  - Kitakyushu
  - Kumamoto
  - Kurume
  - Kyoto
  - Matsumoto
  - Musashino
  - Nagoya
  - Niigata
  - Nishinomiya
  - Ohmura
  - Osaka
  - Ōsaka-sayama
  - Sakai
  - Sapporo
  - Sendai
  - Tokyo
  - Touon
  - Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 17-January-2011 and 22-October-2012 and recruited participants with chronic genotype 1 Hepatitis C Virus (HCV) infection who were treatment-naïve from 37 study centers in Japan. A total 183 participants were randomized and started treatment; 172 completed the study.
Pre-assignment Details: Treatment-naïve HCV-infected participants were assigned to 1 of 2 groups to receive TMC435 100 mg once daily with PegIFN alpha-2a and ribavirin (PR) until Week 12, followed by PR until Week 24 or 48 OR placebo with PR until Week 12, followed by PR until Week 48.
Groups:
- TMC435 100 mg 12 Wks + PR 24/48: Participants were given TMC435 100 mg once daily plus peginterferon alpha-2a (PegIFNα-2a) and ribavirin (RBV) for 12 Weeks (Wks) followed by PegIFNα-2a (P) and RBV (R) until Week 24 (PR24). Treatment was to be stopped at Week 24 for participants who achieved plasma levels of Hepatitis C virus ribonucleic acid (HCV RNA) < 1.2 log10 IU/mL detectable or undetectable at Week 4 and undetectable HCV RNA at Week 12. Other participants continued PR until Week 48 (PR48).
- PBO 12 Wks + PR 48: Participants were given placebo (PBO) once daily plus peginterferon alfa-2a (PegIFNα-2a) and ribavirin (RBV) for 12 Weeks (Wks) followed by PegIFNα-2a (P) and RBV (R) until Week 48 (PR 48).
Period: Overall Study
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48
Started | 123 | 60
Completed | 119 | 53
Not Completed | 4 | 7
Not completed — Other | 1 | 1
Not completed — Withdrawal by Subject | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48 | Total
Number analyzed (Participants) | 123 | 60 | 183
Age, Continuous [Median (Full Range); unit: years] | 56 [23 to 69] | 54.5 [30 to 69] | 55 [23 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 36 | 120
  Male | 39 | 24 | 63

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a Sustained Virologic Response at the End of Treatment (EOT) and 12 Weeks After the Last Dose of Treatment (SVR12)
Description: The table below shows the observed percentage of participants with a SVR12 defined as undetectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) at EOT (Week 24 or 48) and at 12 weeks after the last dose of treatment (Week 36 or 60).
Time Frame: EOT (up to Week 24 or 48) and 12 weeks after the EOT (up to Week 36 or 60)
Population: The Full Analysis Set (FAS) consisted of all participants who received at least one dose of study drug during the study except for those who did not meet the major eligibility criteria for the study and participants who did not have efficacy data available after treatment with study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48
Number analyzed (Participants) | 123 | 60
Percentage of participants | 88.6 [83.63 to 94.39] | 61.7 [49.6 to 73.47]
Statistical Analysis 1: Comparison: TMC435 100 mg 12 Wks + PR 24/48 vs PBO 12 Wks + PR 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The p-value was based on the asymptomatic distribution of the generalized Cochran-Mantel-Haenszel (CMH) statistic controlling for stratification factors; The Cochran-Mantel-Haenszel test was adjusted for stratification factors (age and IL28B genotype); (see comment) = 27.5, 95% CI 2-sided [14.38 to 40.56] — The parameter estimated was the difference of stratum adjusted proportion between groups

2. Secondary Outcome: The Percentage of Participants With a Sustained Virologic Response at the End of Treatment (EOT) and 24 Weeks After the Last Dose of Treatment (SVR24)
Description: The table below shows the observed percentage of participants with a SVR24 defined as undetectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) at the end of treatment (EOT, defined as up to Week 24 or 48) and at 24 weeks after the last dose of treatment (up to Week 48 or 72).
Time Frame: EOT (up to Week 24 or 48) and 24 weeks after the after the last dose of treatment (up to Week 48 or 72)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48
Number analyzed (Participants) | 123 | 60
Percentage of participants | 88.6 | 56.7
Statistical Analysis 1: Comparison: TMC435 100 mg 12 Wks + PR 24/48 vs PBO 12 Wks + PR 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The Cochran-Mantel-Haenszel test was adjusted for stratification factors (age and IL28B genotype); (see comment) = 32.6, 95% CI 2-sided [19.75 to 45.40] — The parameter estimated was the difference of stratum adjusted proportion between groups

3. Secondary Outcome: The Percentage of Participants Who Achieved a Greater Than or Equal to 2 log10 IU/mL Drop From Baseline in Plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) at Each Time Point During Treatment and Follow-up
Description: The table below shows the percentage of participants with greater than (>) or equal to (=) 2 log10 IU/mL drop from baseline in plasma levels of HCV RNA at each time point during treatment and post-treatment follow-up (FU).
Time Frame: Day 3, Day 7 and Weeks 2, 3, 4, 8, 12, 16, 20, 24, 28, 36, 42, 48, 52, 60, 72, EOT (up to Week 24 or 48), FU Week 4, 12, and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48
Number analyzed (Participants) | 123 | 60
Percentage of participants
  Day 3 | 98.4 | 26.7
  Day 7 | 99.2 | 46.7
  Week 2 | 100.0 | 58.3
  Week 3 | 100.0 | 71.7
  Week 4 | 99.2 | 76.7
  Week 8 | 100.0 | 88.3
  Week 12 | 97.6 | 88.3
  Week 16 | 95.1 | 88.3
  Week 20 | 95.9 | 86.7
  Week 24 | 92.7 | 83.3
  Week 28 | 94.3 | 80.0
  Week 36 | 87.8 | 80.0
  Week 42 | 2.4 | 76.7
  Week 48 | 86.2 | 75.0
  Week 52 | 0.0 | 71.7
  Week 60 | 88.6 | 65.0
  Week 72 | 88.6 | 58.3
  EOT (up to Week 24 or 48) | 99.2 | 96.7
  FU Week 4 | 96.7 | 83.3
  FU Week 12 | 89.4 | 65.0
  FU Week 24 | 88.6 | 58.3

4. Secondary Outcome: The Percentage of Participants With Undetectable Plasma Levels of Hepatitis C Virus Ribonucleic Acid (HCV RNA) During Treatment and at the End of Treatment (EOT)
Description: The table below shows the percentage of participants with undetectable plasma levels of HCV RNA <1.2 log10 IU/mL during treatment at Weeks 4, 12, 24, 36, 48, 60, 72, and at the EOT (up to Week 24 or 48).
Time Frame: Weeks 4, 12, 24, 36, 48, 60, 72, and at EOT (up to Week 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48
Number analyzed (Participants) | 123 | 60
Percentage of participants
  Week 4 | 83.7 | 13.3
  Week 12 | 96.7 | 63.3
  Week 24 | 91.9 | 73.3
  Week 36 | 87.0 | 71.7
  Week 48 | 86.2 | 75.0
  Week 60 | 88.6 | 61.7
  Week 72 | 88.6 | 56.7
  EOT (up to Week 24 or 48) | 99.2 | 88.3

5. Secondary Outcome: The Number of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as a confirmed increase of > 1 log10 IU/mL in plasma levels of hepatitis C virus (HCV) ribonucleic acid (RNA)l from the lowest level reached or a confirmed value of plasma HCV RNA of > 2.0 log10 IU/mL in participants whose plasma HCV RNA level had previously been below 1.2 log10 IU/mL detectable or undetectable during the treatment period (up to the end of treatment [EOT]).
Time Frame: Up to EOT (up to Week 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48
Number analyzed (Participants) | 123 | 60
Participants | 1 | 2

6. Secondary Outcome: The Number of Participants Demonstrating Viral Relapse
Description: The table below shows the number of participants who demonstrated viral relapse, defined as undetectable plasma levels of hepatitis C virus (HCV) ribonucleic acid (RNA) at the End of Treatment (EOT) (up to Week 24 or 48) and detectable HCV RNA during follow-up or detectable plasma levels of HCV RNA at the time points of sustained virologic response (SVR) assessment. The incidence of viral relapse was only calculated for participants with undetectable plasma levels of HCV RNA at the EOT and with at least one follow-up HCV RNA. measurement.
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48
Number analyzed (Participants) | 118 | 49
Participants | 9 | 15

7. Secondary Outcome: The Number of Participants With Abnormal Alanine Aminotransferase (ALT) Levels at Baseline Who Achieved Normal ALT Levels at the End of Treatment (EOT)
Description: The table below shows the number of participants with abnormal ALT levels at Baseline (Day 1) who achieved normal ALT levels at the EOT (up to Week 24 or 48). At Baseline, 61/123 participants in the TMC435 treatment group and 25/60 participants in the Placebo treatment group had abnormal ALT levels. At the EOT, 47 (77.0%) participants in the TMC435 treatment group and 18 (72.0%) participants in the Placebo treatment group had ALT levels that returned to normal (or normalization of ALT levels defined as an ALT value less than or equal to the Upper Limit of Normality [ie, 40 IU/mL] at EOT.).
Time Frame: Baseline (Day 1) to EOT (up to Week 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48
Number analyzed (Participants) | 61 | 25
Participants | 47 | 18

8. Secondary Outcome: The Percentage of Participants in the TMC435 Treatment Group Who Met Response Guided Treatment (RGT) Criteria and Completed Treatment With Peginterferon Alpha-2a (PegIFN Alpha-2a) and Ribavirin (RBV) at Week 24
Description: The table below shows the percentage of participants in the TMC435 treatment group who met RGT criteria (ie, who had plasma levels of hepatitis C virus ribonucleic acid [HCV RNA] <1.2 log10 IU/mL detectable/undetectable at Week 4 and <1.2 log 10 IU/mL undetectable at Week 12) and completed treatment with pegIFN alpha 2a and RBV at Week 24. Participants in the TMC435 treatment group not meeting RGT criteria and participants in the placebo group continued treatment with PegIFN alpha 2a and RBV to Week 48.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48
Number analyzed (Participants) | 123
Percentage of participants | 91.9

9. Secondary Outcome: Plasma Concentrations of TMC435
Description: The table below shows median (range) predose plasma concentration (C0h) values and median (range) maximum plasma concentration (Cmax) values for TMC435 for all participants in the TMC435 treatment group. The time frame of "Overall" (up to Week 12) represents the median exposure estimate using all available data for each participant in the study.
Time Frame: Overall (ie, Up to Week 12)
Population: Pharmacokinetic (PK) analysis was performed in the PK population defined as all participants from whom sparse blood samples were drawn and who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48
Number analyzed (Participants) | 123
ng/mL
  C0h | 1005 [64 to 8543]
  Cmax | 2601 [1317 to 10161]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24h) for TMC435
Description: The table below shows the median (range) AUC24h values for TMC435 for all participants in the TMC435 treatment group who received TMC435 for up to 12 weeks. The time frame of "Overall" (up to Week 12) represents the median exposure estimate using all available data for each participant in the study.
Time Frame: Overall (Up to Week 12)
Population: as for outcome 9
Measure: Median (Full Range); unit: ng.h/mL
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48
Number analyzed (Participants) | 123
ng.h/mL | 42721 [11569 to 225205]

ADVERSE EVENTS:
Time Frame: Up to approximately 52 weeks (includes all serious and other adverse events that newly occurred or worsened after treatment with TMC435, PegIFNα-2b or ribavirin, until the end date of the last study medication intake + 28 days).
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | PBO 12 Wks + PR 48
Serious Adverse Events (participants affected / at risk) | 4/123 | 6/60
Other Adverse Events (participants affected / at risk) | 123/123 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 100 mg 12 Wks + PR 24/48 (N=123) | PBO 12 Wks + PR 48 (N=60)
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 100 mg 12 Wks + PR 24/48 (N=123) | PBO 12 Wks + PR 48 (N=60)
White blood cell count decreased (Investigations) | 78 | 41
Neutrophil count decreased (Investigations) | 69 | 37
Platelet count decreased (Investigations) | 60 | 23
Haemoglobin decreased (Investigations) | 27 | 9
Blood bilirubin increased (Investigations) | 20 | 4
Blood triglycerides increased (Investigations) | 17 | 5
Haematocrit decreased (Investigations) | 16 | 8
Red blood cell count decreased (Investigations) | 13 | 6
Lipase increased (Investigations) | 9 | 1
Weight decreased (Investigations) | 9 | 8
Pyrexia (General disorders) | 75 | 31
Malaise (General disorders) | 52 | 27
Injection site reaction (General disorders) | 22 | 9
Fatigue (General disorders) | 13 | 7
Injection site erythema (General disorders) | 4 | 6
Administration site reaction (General disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 57 | 37
Alopecia (Skin and subcutaneous tissue disorders) | 44 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 35 | 18
Erythema (Skin and subcutaneous tissue disorders) | 17 | 4
Eczema (Skin and subcutaneous tissue disorders) | 10 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 9
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 5
Anaemia (Blood and lymphatic system disorders) | 70 | 36
Neutropenia (Blood and lymphatic system disorders) | 8 | 1
Leukopenia (Blood and lymphatic system disorders) | 7 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3
Stomatitis (Gastrointestinal disorders) | 28 | 12
Diarrhoea (Gastrointestinal disorders) | 20 | 17
Abdominal discomfort (Gastrointestinal disorders) | 16 | 5
Nausea (Gastrointestinal disorders) | 16 | 12
Constipation (Gastrointestinal disorders) | 9 | 5
Vomiting (Gastrointestinal disorders) | 6 | 5
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6
Cheilitis (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Gingivitis (Gastrointestinal disorders) | 2 | 3
Toothache (Gastrointestinal disorders) | 1 | 3
Headache (Nervous system disorders) | 54 | 26
Dysgeusia (Nervous system disorders) | 20 | 8
Dizziness (Nervous system disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 28 | 20
Insomnia (Psychiatric disorders) | 27 | 25
Depression (Psychiatric disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 21 | 17
Gastroenteritis (Infections and infestations) | 1 | 3
Retinal exudates (Eye disorders) | 7 | 2
Retinal haemorrhage (Eye disorders) | 7 | 1
Retinopathy (Eye disorders) | 7 | 5
Dry eye (Eye disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Vertigo (Ear and labyrinth disorders) | 8 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.